CLINICAL TRIAL: NCT03054831
Title: The Effect of General Anesthesia on Pharmacokinetics and Pharmacogenomics of Liquid Oxycodone in Pediatric Surgical Patients
Brief Title: The Effect of General Anesthesia on Pharmacokinetics of Oxycodone in Pediatric
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Patcharee Sriswasdi, Attending Anesthesiologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-P00022355
Record Dates: First submitted 2016-10-06; First posted 2017-02-16 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Liquid Oxycodone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Age 2-5 years-Before GA (Active Comparator): The group will include 25 patients (children 2-5 years old). In this group the children will be randomized to receive 0.1mg/kg of liquid oxycodone via an orogastric tube before the procedure at the beginning of general anesthesia (after intubation).
  Interventions: Drug: liquid oxycodone
- Age 2-5 years-After GA (Active Comparator): In this group 25 children will be randomized to receive 0.1mg/kg of liquid oxycodone via an orogastric tube after the procedure at the end of general anesthesia (before extubation).
  Interventions: Drug: liquid oxycodone
- Age 6-8 years-Before GA (Active Comparator): The group will include 25 patients (children 6-8 years old). In this group the children will be randomize to receive 0.1 mg/kg of liquid oxycodone orally before the surgery in pre-op holding.
  Interventions: Drug: liquid oxycodone
- Age 6-8 years-After GA (Active Comparator): The group will include 25 patients (children 6-8 years old). In this group the children will be randomize to receive 0.1 mg/kg of liquid oxycodone orally after surgery in the Post Anesthesia Care Unit (PACU).
  Interventions: Drug: liquid oxycodone

INTERVENTIONS:
Drug: liquid oxycodone — The group will include 25 patients (children 2-5 years old). In this group the children will be randomized to receive 0.1mg/kg of liquid oxycodone via an orogastric tube before the procedure at the beginning of general anesthesia (after intubation).
  In this group 25 children will be randomized to receive 0.1mg/kg of liquid oxycodone via an orogastric tube after the procedure at the end of general anesthesia (before extubation).
  The group will include 25 patients (children 6-8 years old). In this group the children will be randomize to receive 0.1 mg/kg of liquid oxycodone orally before the surgery in pre-op holding.
  The group will include 25 patients (children 6-8 years old). In this group the children will be randomize to receive 0.1 mg/kg of liquid oxycodone orally after surgery in the Post Anesthesia Care Unit (PACU).

SUMMARY:
Oxycodone is an oral opioid analgesic that is most commonly prescribed for the management of pain in post-operative patients at Boston Children's Hospital. Oxycodone has been widely used in adults and children to relieve post-operative pain. However, its pharmacokinetics (what it does in the body) and pharmacodynamics (how it works) have not been well established in children. Some children, because of their specific genetic make-up, may metabolize the drug more quickly and therefore may be at risk for more side effects in the commonly prescribed dose. The investigators would like to find out more about how general anesthesia (GA) effects how this drug is absorbed, metabolized and excreted in children. In order to study these aspects, the investigators would like to give oxycodone to surgical patients (group one will receive oxycodone at the beginning of GA and group two will receive oxycodone at the end of GA) at Boston Children's Hospital then measure its metabolic activity and also perform a specific genetic analysis.

DETAILED DESCRIPTION:
This research will involve two treatment groups: (children 2-5 years old) and (children 6-8 years old). The first group will include 20 children 2-5 years old. In this group the children will be randomized to either receive 0.1mg/kg of liquid oxycodone via an orogastric (OG) tube after induction but before the procedure at the beginning of general anesthesia, or 0.1mg/kg of liquid oxycodone via an OG tube after the procedure at the end of general anesthesia. Every patient will receive inhalational or intravenous induction of anesthesia as decided by the anesthesia team on the day of surgery, as is routine clinical care. An intravenous cannula (IV) will be inserted in every patient as part of their routine clinical care. No additional intravenous line will be required for this study. An arterial line will only be used if indicated by surgical procedure. As part of the study protocol, a blood sample (5 mL) will be taken from the IV and sent for genetic analysis. The genetic testing is specifically to analyze the following genotypes only: cytochrome P450 (CYP) 2D6 and 3A4, which represent the differences in cytochrome P450 metabolism of oxycodone. An orogastric tube will be placed in the stomach (placement verified by routine accepted clinical guidelines) under anesthesia as is part of standard routine clinical care to remove gastric contents. The same orogastric tube will be used for intragastric liquid oxycodone administration in a dose of 0.1 mg/kg either before the procedure (beginning of general anesthesia) or after the procedure (end of general anesthesia). This weight-adjusted dose of 0.1 mg/kg is administered as per standard clinical dosing guidelines at Boston Children's Hospital..

The second group will include 20 patients (children 6-8 years old). In this group the children will be randomize to either receive 0.1 mg/kg of liquid oxycodone per oral (PO) before the surgery in pre-op holding, or 0.1 mg/kg of liquid oxycodone PO after surgery in the Post Anesthesia Care Unit (PACU).

As part of routine clinical care, the anesthesiologist may give any of the following narcotics for additional pain management based on their clinical judgment: Fentanyl, sufentanil, and remifentanyl. For the purposes of this study, the following narcotics will not be administered: morphine and hydromorphone. Additionally, oxycodone will not be administered after the initial study dose in the operating room. These medications produce metabolites that would interfere with the pharmacokinetics being studied. Furthermore, morphine, hydromorphone and oxycodone will be withheld during the entire study period (up to 24 hours). This is not standard clinical care, but withholding morphine/hydromorphone/oxycodone will not result in any additional risk for the patient, since there are equally effective pain management options available which are standard of care. If the clinician deems that morphine, hydromorphone, or oxycodone is necessary for clinical care, it will not be withheld, and the patient will be withdrawn from the study.

A total of 11 blood samples will be drawn for the study. The first sample will be sent for genetic testing. The other 10 samples will be drawn at the following time points: sample 1: within 2 hours of post dose oxycodone, sample 2-7: within 30 to 90 min after last sample drawn and within 12 hours post dose oxycodone, sample 8-10: anytime between 12 to 24 hours post dose oxycodone (assigned as clinically indicated based on duration of surgery to minimize patient disturbance). Therefore, blood samples (1 mL each) will be drawn at 10 different time points in each patient. Blood for the study purposes will be drawn from the existing intravenous line or arterial line at the specific time points indicated when the child is under anesthesia. Postoperatively, regarding the timing of the blood draws, it is not necessary to be exact but rather to accurately record the time that the sample is taken. Thus, this will be coordinated with the drawing of routine laboratory tests if possible, in order to minimize patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

All patients are scheduled for the following in-patient surgical procedures:

* hypospadias repair
* ureteral reimplantation
* pyeloplasty (Genitourinary Surgery Service) and age between 2-8 years, and opioid naive, and not meet exclusion criteria

Exclusion Criteria:

* currently taking cytochrome P450(CYP) 3A4 or 2D6 inhibitors/inducers
* known history of allergy to oxycodone
* known gastrointestinal, hepatic, or renal dysfunction
* known sleep apnea or impaired respiratory reserve
* speak a language other than English

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the effect of general anesthesia on plasma oxycodone level in patients age 2-5 years . | upto 24 weeks
  Plasma oxycodone levels, at 10 time points, will be used to determine the area under the curve(AUC)
the effect of general anesthesia on plasma oxycodone level in patients age 6-8 years | up to 24 weeks
  Plasma oxycodone levels, at 10 time points, will be used to determine the area under the curve(AUC)

SECONDARY OUTCOMES:
the effect of general anesthesia on plasma oxymorphone level in patients age 2-5 years | up to 2 years
  Plasma oxymorphone levels, at 10 time points, will be used to determine the area under the curve(AUC)
the effect of general anesthesia on plasma noroxymorphone in patients age 2-5 years | up to 2 years
  Plasma noroxymorphone levels, at 10 time points, will be used to determine area under the curve(AUC)
the effect of general anesthesia on plasma noroxycodone level in patients age 2-5 years | up to 24 weeks
  Plasma noroxycodone levels, at 10 time points, will be used to determine the area under the curve(AUC)
the effect of general anesthesia on plasma oxymorphone level in patients age 6-8 years | up to 24 weeks
  Plasma oxymorphone levels, at 10 time points, will be used to determine the area under the curve(AUC)
the effect of general anesthesia on plasma noroxymorphone in patients age 6-8 years | up to 24 weeks
  Plasma noroxymorphone levels, at 10 time points, will be used to determine area under the curve(AUC)
the effect of general anesthesia on plasma noroxycodone level in patients age 6-8 years | up to 24 weeks
  Plasma noroxycodone levels, at 10 time points, will be used to determine the area under the curve(AUC)
the effect of general anesthesia on plasma oxycodone level in patients age 2-5 years with respect to the pharmacogenomics. | up to 24 weeks
  Plasma oxycodone levels, at 10 time points, will be used to determine the area under the curve(AUC).
the effect of general anesthesia on plasma oxycodone level in patients age 6-8 years years with respect to the pharmacogenomics. | up to 24 weeks
  Plasma oxycodone levels, at 10 time points, will be used to determine the area under the curve(AUC).
the effect of general anesthesia on oxycodone absorption in patients age 2-5 years | up to 24 weeks
  Plasma oxycodone levels, at 10 time points, will be used to determine the onset of oxycodone absoprtion
the effect of general anesthesia on oxycodone absorption in patients age 6-8 years | up to 24 weeks
  Plasma oxycodone levels, at 10 time points, will be used to determine the onset of oxycodone absoprtion
the effect of general anesthesia on maximum plasma oxycodone level in patients age 2-5 years | up to 24 weeks
  Plasma oxycodone levels, at 10 time points, will be used to determine maximum plasma concentration (Cmax).
the effect of general anesthesia on maximum plasma oxycodone level in patients age 6-8 years | up to 24 weeks
  Plasma oxycodone levels, at 10 time points, will be used to determine maximum plasma concentration (Cmax).

CONTACTS AND LOCATIONS:
Overall Officials: Patcharee Sriswasdi, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes